CLINICAL TRIAL: NCT02700087
Title: In Infants With Symptoms of Tracheomalacia or Laryngomalacia, Does Acid-Blocking Medication Improve Respiratory Symptoms? A Randomized, Controlled Trial
Brief Title: In Infants With Laryngomalacia, Does Acid-Blocking Medication Improve Respiratory Symptoms?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Douglas Sidell, Assistant Professor - Med Center Line, Otolaryngology- Head and Neck Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-35551
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Laryngomalacia; Acid Reflux; Stridor
Keywords: Laryngomalacia
MeSH Terms: conditions — Laryngomalacia; Gastroesophageal Reflux; Respiratory Sounds | interventions — Ranitidine; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- H2 blocker versus placebo (Placebo Comparator): The patient will then be randomly placed in the control group (placebo) or the intervention group (ranitidine 2mg/kg every 12 hours or famotidine 0.5 mg/kg daily).
  Patients will stay on medication for a minimum of 6 months, or until symptoms resolve. Patients will be seen in follow up at 1, 2, 3, 4, 5, 6, 8 and 10 months. At which time I-GERQ, ASQ and weights will be taken. The primary outcome measure will be the time for the ASQ score to drop to normal on ranitidine or famotidine versus placebo.
  Interventions: Drug: ranitidine or famotidine; Drug: Placebo
- Treatment arm (Active Comparator): Patients who develop severe airway symptoms while they are in the H2 blocker versus placebo arm will then cross over to the treatment arm of the study. These patients will exit randomization and be unblinded. These patients will all be given H2 blockers, and the effects of the H2 blockers will be monitored and studied. Alternatively, patients' families may also elect to undergo surgery to treat laryngomalacia.
  Interventions: Drug: ranitidine or famotidine

INTERVENTIONS:
Drug: ranitidine or famotidine — Patients with symptomatic laryngomalacia will receive ranitidine, famotidine, or placebo medications in order to see if these medications help their symptoms to resolve.
Drug: Placebo — Patients with symptomatic laryngomalacia who meet inclusion criteria will be randomized to receive placebo, ranitidine or famotidine, in order to see if these medications help their symptoms to resolve.
  Arms: H2 blocker versus placebo

SUMMARY:
All neonates, ages 0 to 4 months, presenting to LPCH pediatric ENT clinic for airway difficulties or stridor will be screened for inclusion. As is consistent with an acceptable standard of medical care, these children will undergo a flexible nasal endoscopic exam to make the diagnosis of laryngomalacia, as well as be weighed and a breastfeeding history taken. If laryngomalacia is present, the study staff with then administer the Infant Gastroesophageal Reflux Questionnaire (IGERQ) and an airway symptoms questionnaire (ASQ).

Those babies with an IGERQ score of less than sixteen (no more than mild reflux) and an ASQ score greater than six will be eligible for randomization. The patient will then be randomly placed in the control group (placebo) or the intervention group (ranitidine 2mg/kg every 12 hours or famotidine 0.5 mg/kg daily). Patients will stay on medication for a minimum of 6 months, or until symptoms resolve. Patients will be seen in follow up at 1, 2, 3, 4, 5, 6, 8 and 10 months. At which time I-GERQ, ASQ and weights will be taken. The primary outcome measure will be the time for the ASQ score to drop to normal on ranitidine or famotidine versus placebo.

A secondary outcome will be weight gain in percentile. If the patient's I-GERQ score goes above 16 at any time in the study, the patient will be crossed over to the treatment arm and started on medical treatment.

DETAILED DESCRIPTION:
Laryngomalacia, or a soft, floppy upper airway, is the most common cause of noisy breathing in neonates. It is caused by a combination of factors including neuromuscular weakness, cartilaginous inadequacy, and anatomic abnormalities in the voice box. The majority of affected babies' symptoms resolve by one year without intervention, but around 5% of cases require surgical intervention to treat failure to thrive or obstructive sleep apnea.

Many babies with laryngomalacia are treated empirically with H2 blockers such as ranitidine or famotidine to prevent reflux of stomach acid from causing further inflammation in an already compromised upper airway. However, to date no study has been performed to show a definitive benefit of these medications.

The investigators hope to determine whether H2 blockers such as ranitidine and famotidine improve airway symptoms in babies with laryngomalacia. This will have an effect on practice guideline for one of the most common problems encountered in pediatric otolaryngology.

All neonates, ages 0 to 4 months, presenting to LPCH pediatric ENT clinic for airway difficulties or stridor will be screened for inclusion. As is consistent with an acceptable standard of medical care, these children will undergo a flexible nasal endoscopic exam to make the diagnosis of laryngomalacia, as well as be weighed and a breastfeeding history taken. If laryngomalacia is present, the study staff with then administer the Infant Gastroesophageal Reflux Questionnaire (IGERQ) and an airway symptoms questionnaire (ASQ).

Those babies with an IGERQ score of less than sixteen (no more than mild reflux) and an ASQ score greater than six will be eligible for randomization. The patient will then be randomly placed in the control group (placebo) or the intervention group (ranitidine 2mg/kg every 12 hours or famotidine 0.5 mg/kg daily). Patients will stay on medication for a minimum of 6 months, or until symptoms resolve. Patients will be seen in follow up at 1, 2, 3, 4, 5, 6, 8 and 10 months. At which time I-GERQ, ASQ and weights will be taken. The primary outcome measure will be the time for the ASQ score to drop to normal on ranitidine or famotidine versus placebo.

A secondary outcome will be weight gain in percentile. If the patient's I-GERQ score goes above 16 at any time in the study, the patient will be crossed over to the treatment arm and started on medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 0 - 4 months old
* stridor and flexible laryngoscopy demonstrating laryngomalacia
* airway symptom score over 4
* only has physiologic GER (I-GERQ < 16)

Exclusion Criteria:

* requiring surgery for LGM
* other airway dz seen on flexible laryngoscopy
* history of or already on PPI therapy
* minimal/mild airway symptoms (airway score < 4)
* pathologic GERD (I-GERQ greater than 16) - These pts cannot be randomized because this is the standard score in Pediatric GI literature strongly indicating anti-reflux meds
* premature birth (< 36 weeks)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Time to normalization of airway symptoms score | 10 months
  The primary outcome measure will be the time for the ASQ score to drop to normal on ranitidine or famotidine versus placebo.

SECONDARY OUTCOMES:
Weight gain | 10 month
  A secondary outcome will be weight gain in percentile.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Sidell, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson DM. Abnormal sensorimotor integrative function of the larynx in congenital laryngomalacia: a new theory of etiology. Laryngoscope. 2007 Jun;117(6 Pt 2 Suppl 114):1-33. doi: 10.1097/MLG.0b013e31804a5750. PMID 17513991
- [Background] Olney DR, Greinwald JH Jr, Smith RJ, Bauman NM. Laryngomalacia and its treatment. Laryngoscope. 1999 Nov;109(11):1770-5. doi: 10.1097/00005537-199911000-00009. PMID 10569405
- Available data/document: Informed Consent Form: Consent form cycle 3 — https://eprotocol.stanford.edu/irb/ControlServlet?updateFlag=Y